CLINICAL TRIAL: NCT02151942
Title: Patient-Specific Simulation Used for Case Rehearsal Prior to EVAR Procedure - Evaluation of Clinical Performance With and Without Prior Rehearsal Using the Procedure Rehearsal Studio. Multi-center Randomized Study
Brief Title: Patient-Specific Simulation Used for EVAR Procedure Rehearsal - Evaluation of Clinical Performance With and Without Prior Rehearsal
Acronym: PRS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Simbionix US Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PRS-001
Record Dates: First submitted 2014-05-21; First posted 2014-06-02 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Infra Renal Aortic Aneurysm
Keywords: elective endovascular AAA repair

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Procedure/Surgery : Endovascular Aneurysm Repair with no prior procedure rehearsal
- Rehearsal group: Procedure/Surgery : Endovascular Aneurysm Repair with prior procedure rehearsal

SUMMARY:
The purpose of this study is to evaluate the procedural and clinical benefits of patient specific pre-procedure rehearsal for operators with various experience levels as a tool for optimizing Endovascular Aneurysm Repair (EVAR) procedures.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Elective patients planned to undergo EVAR procedures with an endograft compatible with the Simbionix PRS.
3. Computed Tomography Angiography (CTA) scan of the abdominal aorta performed as standard of care. Sufficient quality/defined protocol.

Exclusion Criteria:

1. Subject is below 18 years old
2. Operator cannot complete the indicated rehearsal and practice.
3. Patients requiring emergent aneurysm treatment, e.g. trauma or rupture.
4. Arterial dissection.
5. Patients with Stage 4 of chronic kidney disease (GFR<30 ml/min/m2).
6. Patient is indicated for use of snorkels, chimneys, fenestrated or branched graft devices
7. Pregnant or lactating women.
8. Off label stent graft use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted for elective endovascular AAA repair will be randomized
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Overall Fluoro time | Within 4 hr. after EVAR procedure starts
Subjective operator perceived effectiveness of prior procedure rehearsal | Within 4 hr. after EVAR procedure starts

SECONDARY OUTCOMES:
Intraprocedural safety measurements | Within 4 hr. after EVAR procedure starts
  1. Overall contrast use (volume)
  2. Skin entry radiation dose
  3. Overall procedure time (from gaining bilateral access until the satisfactory completion of endograft deployment, excluding all adjunctive procedures such as hypogastric embolization, Iliac Percutaneous Transluminal Angioplasty (PTA)/Stenting, sheath removal and hemostasis time)
  4. Procedural blood loss - number of transfused units
  5. Arterial injury (dissection, perforation, rupture, surgical conversion, embolization, none)
Change in procedure plan | Within 4 hr. after EVAR procedure rehearsal starts
  Comparison of treatment plans based on Customary (normal institutional) technique, following 3D reconstruction, and after simulation procedures.
Adjunctive device utilization | Within 4 hr. after EVAR procedure ends
  Number and type of used wires, catheters, stent grafts, additional stent graft components and balloons
Gate cannulation time | Within 3 hr. after EVAR procedure starts
  Time to cannulate the contralateral gate with a wire.
Similarity of simulation to actual case | Within 3 hr. after EVAR procedure ends
  1. Anatomy
  2. Anticipated devices (sizing, tools)
  3. Fluoroscopic Angulations
  4. Case complexity
General satisfaction- Subjective experience of simulation experience | Within 4 hr. after EVAR procedure ends
  1. Overall ease of use
  2. Controls
  3. Imaging
  4. Device exchanges
  5. Device performance
Cost analysis | Within the first 30 days after the EVAR procedure
Technical/Clinical success rate | Within the first 30 days after the EVAR procedure
  Successful endograft deployment and absence of type 1 or 3 endoleak
Time of simulator rehearsal | Within 3 hr. after EVAR procedure rehearsal ends
Time in ICU | within 30 days after the EVAR procedure
Overall Length of Stay | Within 30 days after the EVAR procedure

CONTACTS AND LOCATIONS:
Overall Officials: John H. Rundback, MD, Principal Investigator — Holy Name Medical Center
Locations (7):
- United States (5):
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - University of South Florida, Tampa General Hospital, Tampa, Florida
  - Holy Name Medical Center, Teaneck, New Jersey
  - University Hospital Case Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
- C.H.U De Nancy, Nancy, France
- Policlinico S. Orsola-Malpighi, Bologna, Italy